CLINICAL TRIAL: NCT00425568
Title: Phase I Study of Transdermal Testosterone Gel and Its Effect on Erection Quality as Measured by a Digital Inflection Rigidometer (DIR)
Brief Title: Transdermal Testosterone Gel/Effect on Erection Quality as Measured by DIR
Status: Completed | Type: Observational
Sponsor: Lamm, Steven, M.D. (Individual)
Collaborators: Solvay Pharmaceuticals (Industry)
Other Study IDs: DIR1-SLGSC
Record Dates: First submitted 2007-01-20; First posted 2007-01-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2007-12

CONDITIONS: Hypogonadism
Keywords: hypogonadism; low testosterone level; gonadal deficiency
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: AndroGel (Transdermal Testosterone Gel)

SUMMARY:
Low testosterone may be responsible for "soft" erections in men. The purpose of our study is to see whether the daily application of a testosterone gel to raise testosterone levels will also increase the "hardness" of a man's erection.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone <350 ng/dL,
* 21-59 years of age,
* BMI <30

Exclusion Criteria:

* Those with carcinoma of the breast or known or suspected carcinoma of the prostate or with known hypersensitivity to any of the ingredients in AndroGel.
* Men will be excluded if they have unstable angina, hypertension, diabetes, heart failure, or coronary artery disease.
* Men will agree to discontinue use of current testosterone replacement, as well as Viagra or any other PDE5 inhibitors for 30 days.

Ages: 21 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lamm, M.D., Principal Investigator
Locations (1):
- Steven Lamm, M.D., New York, New York, United States